CLINICAL TRIAL: NCT02659709
Title: Interest of Patients and Their Caregivers in A Smartphone- and Tablet-Based Application for Patients With Glaucoma
Brief Title: Interest in Electronic Applications for Patients With Glaucoma
Acronym: GlaucomaApp
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Jonathon Myers, Principal Investigator, Wills Eye
Other Study IDs: 14-413E
Record Dates: First submitted 2015-08-06; First posted 2016-01-20 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Smartphone; Tablet; Application; Eye Drops
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glaucoma Patients and Caregivers: Glaucoma patients and caregivers will complete a 20 item questionnaire providing demographic information, glaucoma eye drop compliance, interest in medication reminders, availability to smartphone, tablet and social media technology and interest in using a glaucoma application on social media.
  Interventions: Device: Interest in medical education through social media

INTERVENTIONS:
Device: Interest in medical education through social media — Measuring interest in social media technology designed to educate glaucoma patients about disease, testing, and treatments with reminders for taking medications.
  Other Names: Glaucoma App Interest

SUMMARY:
To evaluation interest in use of smartphone- and tablet-based application (app) for participants with glaucoma, ocular hypertension, those at risk and their caregivers.

DETAILED DESCRIPTION:
This study is designed to determine the amount of interest in an educational application (app) on social media for glaucoma patients and their caregivers.

The purpose of this App is to enhance understanding of glaucoma by using short video tutorials. The App will include glaucoma eye drop medication reminders, a short video tutorial which aims to improve understanding of how visual field testing should be performed, how to administer eye drops and a feature that will enable participants to store and organize testing results using a mobile device.

ELIGIBILITY:
Inclusion Criteria:

* Anyone affected by glaucoma
* Family and friends of someone with glaucoma

Exclusion Criteria:

* unable to complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients or care givers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Myers, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Waisbourd M, Dhami H, Zhou C, Hsieh M, Abichandani P, Pro MJ, Moster MR, Katz LJ, Hark LA, Myers JS. The Wills Eye Glaucoma App: Interest of Patients and Their Caregivers in a Smartphone-based and Tablet-based Glaucoma Application. J Glaucoma. 2016 Sep;25(9):e787-91. doi: 10.1097/IJG.0000000000000504. PMID 27552513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Glaucoma patients and Caregivers were recruited from the Glaucoma Service at Wills Eye Hospital, Philadelphia, PA, USA.
Groups:
- Glaucoma Patients and Caregivers: Glaucoma patients and caregivers will test a glaucoma smartphone application (app) on smart phones or tablets then complete 20 item questionnaire providing demographic information, effectiveness and ease of use with the application designed to educate glaucoma patients about disease, testing, and treatments with reminders for taking medications.
Period: Overall Study
Arm/Group | Glaucoma Patients and Caregivers
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fifty participants agreed to answer questions in the survey.
Groups:
- Glaucoma Patients and Caregivers: 50 Glaucoma patients and/or caregivers will test a glaucoma application (app) on smart phones or tablets then complete a 20 item questionnaire providing demographic information, effectiveness and ease of use with the application designed to educate glaucoma patients about disease, testing, and treatments with reminders for taking medications.
Arm/Group | Glaucoma Patients and Caregivers
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 32
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 33
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Patients Owning Smartphone/Tablet Technology
Description: Responses collected from participants about owning access to social media via smartphone or tablet technology obtained by completing a 20 item questionnaire.
Time Frame: 1 hour
Population: Participants responding Yes to owning a smartphone or tablet.
Measure: Count of Participants; unit: Participants
Groups:
- Glaucoma Smartphone Application: Glaucoma patients and/or caregivers answered a Questionnaire on availability to Smartphone or Tablet Usage and accessing social media. Questionnaire includes 20 items regarding demographic information, effectiveness of social media and compliance with glaucoma medications.
  From this information, Smartphone Application will be designed to educate glaucoma patients about the disease, testing, and treatments and also include reminders for taking medications.
Arm/Group | Glaucoma Smartphone Application
Number analyzed (Participants) | 50
Participants | 34

2. Primary Outcome: Patients Having Access to Social Media Via Smartphone or Tablet in the Home
Description: Responses collected from participants about their personal access, through other members in the home, to social media via smartphone or tablet technology obtained by completing a 20 item questionnaire.
Time Frame: 1 hour
Population: Participants responding Yes to anyone in the house owning a smartphone or tablet.
Measure: Count of Participants; unit: Participants
Arm/Group | Glaucoma Smartphone Application
Number analyzed (Participants) | 50
Participants | 39

3. Secondary Outcome: Glaucoma Medication Compliance
Description: Responses collected from participants about compliance to using their glaucoma drops as prescribed obtained by completing a 20 item questionnaire.
Time Frame: 1 hour
Population: Participants responding Yes using their glaucoma eye drops as prescribed.
Measure: Count of Participants; unit: Participants
Arm/Group | Glaucoma Smartphone Application
Number analyzed (Participants) | 50
Participants | 25

4. Secondary Outcome: Use of Medication Reminder
Description: Responses collected from participants about use of medication reminders for their glaucoma drops obtained by completing a 20 item questionnaire.
Time Frame: 1 hour
Population: Participants responding Yes to using their glaucoma eye drops as prescribed without reminders.
Measure: Count of Participants; unit: Participants
Arm/Group | Glaucoma Smartphone Application
Number analyzed (Participants) | 50
Participants | 28

ADVERSE EVENTS:
Time Frame: 1 hour
Groups:
- Glaucoma Smartphone Application: 50 Glaucoma patients and caregivers will test a glaucoma smartphone application (app) on smart phones or tablets then complete 20 item questionnaire providing demographic information, effectiveness and ease of use with the application.
  Smartphone Application: Smartphone Application designed to educate glaucoma patients about disease, testing, and treatments with reminders for taking medications.
Arm/Group | Glaucoma Smartphone Application
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
Participants were recruited from single urban eye care hospital. Results did not distinguish between glaucoma patients and caregivers. Participation did not include testing of the application.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No